CLINICAL TRIAL: NCT06606847
Title: A Phase II, Open-label, Multicentre, Single-arm Study of Durvalumab Plus Oleclumab in Patients With Locally Advanced, Unresectable Non-small Cell Lung Cancer Who Have Not Progressed Following Definitive, Platinum-Based Chemoradiation Therapy (LADOGA)
Brief Title: A Study to Investigate the Effects of Durvalumab With Oleclumab Following Chemoradiation in Participants With Locally Advanced Unresectable Non-Small Cell Lung Cancer (LADOGA)
Acronym: LADOGA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZ-RU-00003
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Locally Advanced NSCLC; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Antineoplastic Agents, Immunological; Antineoplastic Agents; Durvalumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Lung Neoplasms | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: All participants will receive durvalumab and oleclumab as an IV infusions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): durvalumab plus oleclumab as an IV infusions
  Interventions: Drug: Oleclumab; Drug: Durvalumab

INTERVENTIONS:
Drug: Oleclumab — Oleclumab IV (intravenous infusion)
Drug: Durvalumab — Durvalumab IV (intravenous infusion)

SUMMARY:
The purpose of this Phase II, open-label, multicentre, single-arm study is to assess efficacy and safety of durvalumab (MEDI4736) in combination with oleclumab (MEDI9447) in participants with locally advanced (Stage III), unresectable non-small cell lung cancer (NSCLC), who have not progressed following platinum-based concurrent or sequential chemoradiotherapy (cCRT or sCRT).

DETAILED DESCRIPTION:
This is a Phase II, open-label, multicentre, single-arm study assessing the efficacy and safety of durvalumab in combination with oleclumab in participants with locally advanced (Stage III), unresectable NSCLC with WHO performance status of 0 or 1, who have not progressed on prior platinum-based CRT.

All participants will be assigned to receive durvalumab and oleclumab as an IV infusions for up to 12 months (last dose should be administered at week 48). The last administration at Week 48, or until clinical progression, confirmed RECIST 1.1-defined radiological progression, unacceptable toxicity, withdrawal of consent, or an intervention discontinuation criterion is met.

The results of this study will provide clinical data on efficacy and safety of an innovation treatment in the new region - Russian Federation.

ELIGIBILITY:
INCLUSION CRITERIA:

* Participant must be ≥ 18 years at the time of screening.
* Histologically-documented NSCLC and have been treated with concurrent or sequential CRT for locally advanced, unresectable (Stage III) disease.
* Documented tumour PD-L1 status by qualified lab (local or central).
* Documented EGFR and ALK wild-type status (local or central).
* Patients must not have progressed following definitive, platinum based, concurrent or sequential chemoradiotherapy.
* Participants must have received at least 2 cycles of platinum-based chemotherapy before or concurrent with radiation therapy.
* Participants must have received a total dose of radiation of 60 Gy ±10% (54 Gy to 66 Gy) as part of the chemoradiation therapy, to be enrolled. Radiation therapy should be administered by intensity modulated RT/volumetric modulated arc therapy (preferred) or 3D-conforming technique.
* WHO performance status of 0 or 1.
* Adequate organ and marrow function.

EXCLUSION CRITERIA:

* History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥5 years before the first dose of study intervention and of low potential risk for recurrence, adequately resected non-melanoma skin cancer and curatively treated in situ disease, or adequately treated carcinoma in situ or Ta tumours without evidence of disease.
* Mixed small cell and non-small cell lung cancer histology.
* Participants with locally advanced (Stage III) unresectable NSCLC who have progressed during platinum-based CRT.
* Any unresolved toxicity CTCAE >Grade 2 from the prior chemoradiation therapy (excluding alopecia).
* Participants with ≥grade 2 pneumonitis from prior chemoradiation therapy.
* History of idiopathic pulmonary fibrosis, drug-induced pneumonitis, or idiopathic pneumonitis - regardless of time of onset prior to study treatment assignment. Evidence of active non-CRT induced pneumonitis (≥ Grade 2), active pneumonia, active ILD, active or recently treated pleural effusion, or current pulmonary fibrosis.
* Active or prior documented autoimmune or inflammatory disorders (with exceptions).
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) at 12 months | From date of first dose until 12 months
  PFS12 is defined as the Kaplan-Meier estimate of PFS at 12 months per RECIST 1.1 as assessed by the investigator.

SECONDARY OUTCOMES:
Progression free survival (PFS) at 6, 18, and 24 months | From date of first dose until 24 months
  PFS6, PFS18 and PFS24 are defined as the Kaplan-Meier estimate of PFS at 6 months, 18 months and 24 months respectively, per RECIST 1.1 as assessed by the investigator.
Progression Free Surival (PFS) | Up to 24 months after the last patient's first dose
  PFS is defined as time from the start of treatment until progression per RECIST 1.1 as assessed by the investigator, or death due to any cause.
Overall survival (OS) at 12 and 24 months | From date of first dose until 12 and months, respectively
  OS12 and OS24 are defined as the Kaplan-Meier estimate of OS at 12 months and 24 months respectively
Overall Survival (OS) | Up to 24 months after the last patient's first dose
  OS is defined as time from the start of treatment until the date of death due to any cause
Objective response rate (ORR) | Up to 24 months after the last patient's first dose
  ORR is defined as the proportion of participants who have a confirmed complete response (CR) or partial response (PR), as determined by the investigator per RECIST 1.1
Duration of response (DoR) | Up to 24 months after the last patient's first dose
  DoR is defined as the time from first response until progression per RECIST 1.1 as assessed by the investigator, or death due to any cause
Time to Response (TTR) | Up to 24 months after the last patient's first dose
  TTR is defined as the time from the start of the treatment to the first documented objective tumor response observed for participants who achieved CR or PR, as determined by the investigator according to RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (8):
- Russia (8):
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Obninsk
  - Research Site, Saint Petersburg
  - Research Site, Ufa
  - Research Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home